CLINICAL TRIAL: NCT00785564
Title: Imaging Cardiac Electrical Remodeling With ECGI
Brief Title: Imaging Cardiac Electrical Remodeling With Electrocardiogram Imaging (ECGI)
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 07-0995
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Sick Sinus Syndrome
Keywords: T-wave memory; Sick Sinus Syndrome
MeSH Terms: conditions — Sick Sinus Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A consequence of chronic RV pacing is a process of electrical remodeling that alters myocardial repolarization to reflect the altered depolarization induced by the RV lead. When RV pacing is discontinued, the altered repolarization persists for several weeks. This phenomena is traditionally described as "T-wave memory" based upon the 12-lead ECG appearance of inverted T-Waves. The investigators are using the ECGI technique to produce three dimensional electroanatomical images of this phenomena in patients with dual chamber pacemakers. Echocardiography will also be used to image the mechanical effects of RV pacing and T-wave memory. The images will show the spatial distribution of altered repolarization and allow us to correlate any mechanical consequences of this phenomena that may exist.

ELIGIBILITY:
Inclusion Criteria:

* Implanted dual chamber pacemaker for sick sinus syndrome with no history of complete heart block.

Exclusion Criteria:

* Persistent atrial fibrillation that is not suppressed by medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of a pacemaker clinic
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2007-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
ECGI Image | 1 month after RV pacing

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell N Faddis, MD PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States